CLINICAL TRIAL: NCT01874366
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Safety, Tolerability, Pharmacokinetics, Food Effect and Pharmacodynamics of Single and Multiple Ascending Doses of P11187
Brief Title: Determination of Safety,Tolerability,Pharmacokinetics,Food Effect& Pharmacodynamics of Single & Multiple Doses of P11187
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Piramal Enterprises Limited (Industry)
Collaborators: Quintiles, Inc. (Industry); Miami Research Associates (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P11187/77/13
Record Dates: First submitted 2013-05-17; First posted 2013-06-11 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Overweight; Diabetes Mellitus Type 2 in Obese
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P11187 (Experimental): * Part I: Step wise dose escalation in subsequent cohorts and will be based upon the review of safety and tolerability results of the preceding cohort
  * Part II: Step wise dose escalation in the multiple dosing for 14 consecutive days after review of the safety and tolerability of the preceding cohorts
  * Part III: Study drug will be administered under the fasted or fed conditions in two different periods separated by a wash-out interval of 7-10 days
  Interventions: Drug: P11187
- Placebo (Placebo Comparator): Placebo capsules will be matching in appearance with the active drug capsules of P11187.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P11187 — * Part I: Step wise dose escalation(10 to 1500 mg, qd, Oral)
  * Part II: Step wise dose escalation in multiple dosing (≤ 1500 mg, qd, Oral) for 14 consecutive days.
  * Part III: Study drug administered (≤ 1500 mg, qd, Oral) under fasted or fed conditions in two different periods separated by a wash-out interval.
  Other Names: Oral G-Protein Coupled Receptor 40(GPR40)agonist
  Arms: P11187
Drug: Placebo — Placebo capsules will be matching in appearance with the active drug capsules of P11187.
  * In Part I, there will be up to 6 cohorts of 8 subjects each in single dose assessment. Two subjects from each cohort will be dosed with placebo
  * In Part II, there will be 3 cohorts of 12 subjects each and three subjects from each cohort will be dosed with placebo
  Arms: Placebo

SUMMARY:
* Study to Determine the Safety, Tolerability, Pharmacokinetics, Food Effect and Pharmacodynamics of Single and Multiple Ascending Doses of P11187
* It will be conducted in three parts, as described below:
* Part I will be the Single Ascending Dose (SAD) study
* Part II will be the Multiple Ascending Dose (MAD) study
* Part III will be the food effect evaluation

DETAILED DESCRIPTION:
* In Part I, the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single ascending doses of P11187 will be studied in healthy, overweight or obese, male and females (of non-child bearing potential) subjects. There will be up to 6 cohorts of 8 subjects each. At each dose level, 6 subjects will receive a single dose of active treatment, P11187 and 2 subjects will receive a single dose of matching placebo. It is planned that up to 6 dose levels of P11187 may be evaluated after single dose administration.
* In Part II, the safety, tolerability, PK and PD of multiple ascending doses of P11187 administered once daily for 14 consecutive days will be studied in overweight or obese, male and female of non-child bearing potential subjects with type 2 diabetes mellitus. Up to 3 dose levels of P11187 are planned to be evaluated in 3 cohorts of 12 subjects each for 14 days.At each dose level, 9 subjects will receive the active drug, P11187 and 3 subjects will receive matching placebo, once daily for a period of 14 days.
* In Part III, the food effect evaluation of P11187 will be performed in a randomized, open-label, cross-over, two-period study at a single dose level in a cohort of 12 healthy male subjects to be administered the drug under fasted and fed conditions.Subjects will be administered a single dose of P11187 in Periods 1 and 2 under fasted and fed conditions as per the randomization schedule, with a wash-out interval of 7-10 days between the two periods. Subjects who have received the study drug, P11187 under fasted conditions in Period 1 will cross-over and receive the study drug under fed conditions in Period 2 and vice versa.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing to give written informed consent to participate in the study
2. Male & female subjects aged between 18 &70 years (both inclusive) in Part I & II) & between 18 &70 years (both inclusive) in Part III
3. Subjects with a body mass index (BMI) between 19 &42 kg/m2(Part I), 22 &42 kg/m2 (Part II) & 19 &27 kg/m2 (Part III)
4. Healthy subjects having no clinically significant abnormalities in medical history, physical examination, clinical laboratory tests, vital signs & 12-lead electrocardiograms (ECG)
5. Female subjects of non-child-bearing potential, post-menopausal or surgically sterilized (Part I & II)
6. Male subjects agreed to use contraceptive methods as per protocol during & approximately 30 days after the exit/completion of their participation in the study
7. Part II: Subjects with type 2 diabetes mellitus at least 6 mths prior to screening
8. Part II: Subjects on diet & exercise alone or on a stable dose of metformin for a period of at least 2 mths before screening. Subjects who are washed off other medications such as sulfonyureas /alpha-glucosidase inhibitors, at least 14 days prior to dosing.
9. Part II-Subjects with HbA1c between 6 &11% at screening
10. Part II-Subjects with fasting plasma glucose of ≤ 14.42 mmol/L (~260 mg/dL) at screening
11. Part II-Subjects with C-peptide value of > 0.266 nmol/L (0.8 ng/mL) at screening

Exclusion Criteria:

1. Subjects with history of (H/O) significant gastrointestinal, cardiac, renal or liver impairment
2. Subjects with known congenital QTc prolongation or QTcF greater than 450 ms
3. Subjects with H/O hypo/hyperthyroidism (except replacement with thyroxine & on a stable dose since the past 2 mths), repeated thyroid stimulating hormone (TSH) values that is abnormal at screening or subjects with a H/O obesity of endocrine origin
4. Subjects with H/O anaphylaxis/angioedema, adult bronchial asthma, peptic ulcer & clinically important food/drug allergy
5. Subjects with H/O drug abuse/addiction/use of recreational drugs ,mental handicap, psychiatric disorders including eating disorders/seizures /significant head trauma
6. Subjects with H/O alcoholism for more than 2 years /consumption of more than 3 alcoholic drinks per day/consumption of alcohol, 2 days prior to confinement/ during the study
7. Subjects with prior exposure to P11187/ have participated in previous cohorts or have participated in another clinical trial 30 days prior to screening
8. Subjects undergone weight-loss surgery/ consuming prescription drugs including sedatives &steroids within 30 days before first drug administration/ using over-the-counter drugs including herbal/ health supplements & others such as St. John's Wort extract . Subjects consumed weight loss medications within 90 days before the first drug administration.
9. Part II- Subjects with using insulin within 6 mths prior to screening except when used for short duration (less than 14 days) or was being treated with GLP-1 analogues / other anti-diabetic medications except metformin within 6 mths prior to screening. Subjects being treated with herbal/OTC drugs including sulfonylureas/alpha-glucosidase inhibitors unless discontinued/washed-out at least 14 days prior to dosing.Subjects on anti-hypertensive &lipid-lowering medications (only statins) will only be allowed if they are at the same dose since the past 2 mths & are maintained at the same dose throughout the study duration.
10. Part II-Subjects with H/O metabolic complications, mature Onset Diabetes of the Young (MODY)/insulin-dependent type 2 diabetes mellitus/ other unusual forms of diabetes mellitus. Subjects with known endocrine disorders
11. Part II-Subjects with H/O heart failure (NYHA class III &IV)/myocardial infarction/unstable angina /cerebrovascular accident
12. Part II-Subjects with severe/uncontrolled hypertension(above 160/100 mm Hg)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (single and multiple dose studies) | 12-14 Months
  * The safety and tolerability of single ascending doses of P11187 in healthy, overweight and/or obese, male and non-child bearing female subjects (Part I).
  * The safety and tolerability of multiple ascending doses of P11187 in overweight and/or obese, male and non-child bearing female subjects with type 2 diabetes mellitus (Part II).
Food Effect | 12-14 Months
  The effect of food on the pharmacokinetics (PK) of P11187 following single oral doses in healthy male subjects, under fed and fasted conditions (Part III).

SECONDARY OUTCOMES:
Change in Oral Glucose Tolerance Test (OGTT) | 12-14 month
  To determine the effect of single doses of P11187 on pharmacodynamic (PD) parameters (Part I) in the study population defined as follows:
  * Change in Oral Glucose Tolerance Test (OGTT) variables such as glucose AUC, insulin AUC, C-peptide AUC, glucagon AUC, GLP-1 AUC and GIP AUC.
Area under the plasma concentration (AUC) | 12- 14 Month
  * To characterize the pharmacokinetics of P11187 following single and multiple doses (Part I and Part II) in the study population as defined.
  * A non-compartmental PK method will be used to analyze the plasma levels of P11187 on Days 1 (Part I, II & III) and Day 14 (Part II)
  * The PK profile will be derived from the P11187 plasma concentration data in both periods i.e. fasted and fed states (Part III).
Change in Intravenous Glucose Tolerance Test | 12- 14 Month
  * Multiple doses of P11187 on pharmacodynamic (PD) parameters (Part II) in the study population defined as follows:
  * Change in Intravenous Glucose Tolerance Test (IVGTT) variables including glucose , insulin and C-peptide will be measured following an IVGTT.
Change in the Mixed Meal Tolerance Test | 12- 14 Month
  * To determine the effect of multiple doses of P11187 on pharmacodynamic (PD) parameters (Part II) in the study population defined as follows:
  * Change in the Mixed Meal Tolerance Test (MMTT) variables such as glucose , insulin, C-peptide, glucagon, GLP-1 and GIP.
Peak Plasma concentration (Cmax) | 12- 14 Month
  * To characterize the pharmacokinetics of P11187 following single and multiple doses (Part I and Part II) in the study population as defined.
  * A non-compartmental PK method will be used to analyze the plasma levels of P11187 on Days 1 (Part I, II & III) and Day 14 (Part II)
  * The PK profile will be derived from the P11187 plasma concentration data in both periods i.e. fasted and fed states (Part III).
Time to peak plasma concentration (t-max) | 12- 14 Month
  * To characterize the pharmacokinetics of P11187 following single and multiple doses (Part I and Part II) in the study population as defined.
  * A non-compartmental PK method will be used to analyze the plasma levels of P11187 on Days 1 (Part I, II & III) and Day 14 (Part II)
  * The PK profile will be derived from the P11187 plasma concentration data in both periods i.e. fasted and fed states (Part III).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pardo,, MD, Principal Investigator — Phase I clinic: MRA Clinical Research
Locations (1):
- Phase I clinic: MRA Clinical Research, Miami, Florida, United States